CLINICAL TRIAL: NCT02773888
Title: An Evaluation of Non-Invasive ICP Monitoring in Patients Undergoing Invasive ICP Monitoring Via an Intraparenchymal Pressure Monitoring Device
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment temporarily held for site retraining
Sponsor: HeadSense Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-018
Record Dates: First submitted 2016-05-12; First posted 2016-05-16 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Intracranial Hypertension; Brain Injuries; Stroke; Hydrocephalus; Brain Neoplasms
Keywords: intracranial pressure; noninvasive monitoring
MeSH Terms: conditions — Intracranial Hypertension; Brain Injuries; Stroke; Hydrocephalus; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HS-1000 recording (Experimental): ICP readings will be recorded in parallel from both the invasive ICP monitor, and HeadSense's non-invasive ICP monitor. Each recording session will be done until an aggregate of at least 30 minutes worth of quality data is collected, depending on the patient's clinical condition. For each patient, two recording sessions will be completed for 30-60 minutes each for 120 minutes total.
  Interventions: Device: HS-1000

INTERVENTIONS:
Device: HS-1000

SUMMARY:
Invasive intracranial pressure (ICP) monitoring is highly effective, but involves risks. HS-1000 measures ICP non-invasively by assessing the acoustic properties of the patient's head.

HS-1000 device, a proprietary non-invasive ICP monitor, is expected to safely and accurately monitor ICP with minimal discomfort to patients, and provide information about normal or elevated ICP levels to the physicians.

DETAILED DESCRIPTION:
A prospective study will be conducted on 80 patients with an inserted invasive intraparenchymal ICP monitor. Once a patient undergoes invasive ICP monitoring, has a life expectancy of greater than 48 hours and is 14 years old and over at the screening visit, and has an intact/continuous dura layer, the patient will become a candidate for enrollment into the study. If the patient signs the informed consent or the patient's legal authorized representative signs on the patient's behalf, the patient will be enrolled into the trial. Each enrolled patient will be monitored in parallel to the invasive ICP monitor with the HeadSense's device. Once the data collection is complete, results will be analyzed by comparing ICP readings from both devices.

The primary end-point of the study is to collect 60-120 minutes of ICP monitoring data over two sessions of 30-60 minutes each for 80 neurosurgery patients of any etiology. The secondary endpoint of this study is evaluate the safety of the device as measured by incidence of adverse events and serious adverse events over each subject's 96 hours of participation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, aged 14 years old and over at screening visit
* Patient with invasive ICP monitor due to suspected ICP elevation, regardless of etiology
* Survival expectancy greater than 48 hours
* Subject or legal authorized representative (per local regulation) is able and willing to comply with the requirements of the protocol
* Subject or legal authorized representative (per local regulation) is able to understand and sign written informed consent to participate in the study

Exclusion Criteria:

* Subject with ear disease, ear trauma
* Subject with a punctured or discontinuous dura layer (must be intact)
* Subject with cerebral fluid (CSF) leakage
* Known allergy or hypersensitivity to any of the test materials or contraindication to test materials
* Subjects currently enrolled in or less than 30 days post-participation in other investigational device or drug study(s), or receiving other investigational agent(s)
* Any condition that may jeopardize study participation (e.g., abnormal clinical or laboratory finding) or interpretation of study results, or may impede the ability to obtain informed consent (e.g. mental condition)

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of ICP values obtained by the HS device that correlate to ICP using current standards | 30 minutes

SECONDARY OUTCOMES:
Incidence of adverse events during and after recording sessions | 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Katsuji Shima, Principal Investigator — National Defense Medical College
Locations (5):
- Japan (5):
  - Kuki General Hospital, Saitama
  - National Defense Medical College Hospital, Saitama
  - Juntendo University Shizuoka Hospital, Shizuoka
  - Nippon Medical School, Tokyo
  - Tokyo Jikei University Kashiwa Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No